CLINICAL TRIAL: NCT01999842
Title: An Observer-blind Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine(s) GSK3206641A and GSK3206640A Administered in Adults 18 to 64 Years of Age
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Influenza Vaccine(s) GSK3206641A and GSK3206640A Administered in Adults 18 to 64 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201072
Record Dates: First submitted 2013-11-21; First posted 2013-12-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: H7N9; Influenza; Safety; Adults; Adjuvant; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Formulation 1 Group (Experimental): Subjects in this group will receive two doses of GSK3206641A H7N9 vaccine formulation 1 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3206641A
- Formulation 2 Group (Experimental): Subjects in this group will receive two doses of GSK3206641A H7N9 vaccine formulation 2 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3206641A
- Formulation 3 Group (Experimental): Subjects in this group will receive two doses of GSK3206641A H7N9 vaccine formulation 3 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3206641A
- Formulation 4 Group (Experimental): Subjects in this group will receive two doses of GSK3206641A H7N9 vaccine formulation 4 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3206641A
- Formulation 5 Group (Experimental): Subjects in this group will receive two doses of GSK3206640A H7N9 vaccine formulation 5 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3206640A
- Placebo Group (Placebo Comparator): Subjects in this group will receive two doses of placebo at a 21 day interval
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Investigational H7N9 vaccine GSK3206641A — One dose of GSK3206641A H7N9 vaccine administered intramuscularly (IM) in the deltoid region of arm at Day 0 and the second dose of GSK3206641A H7N9 vaccine administered IM in the deltoid region of arm at Day 21
  Arms: Formulation 1 Group; Formulation 2 Group; Formulation 3 Group; Formulation 4 Group
Biological: Investigational H7N9 vaccine GSK3206640A — One dose of GSK3206640A H7N9 vaccine administered IM at the deltoid region of arm at Day 0 and the second dose of GSK3206640A H7N9 vaccine administered IM at the deltoid region of arm at Day 21
  Arms: Formulation 5 Group
Biological: Placebo — One dose of placebo administered IM at the deltoid region of arm at Day 0 and the second dose of placebo administered IM at the deltoid region of arm at Day 21
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of different formulations of GSK Biologicals' H7N9 influenza vaccine in subjects 18 to 64 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults who are 18 to 64 years of age (inclusive) at the time of first study vaccination.
* Written informed consent obtained from subject.
* Subjects who the investigator believes can and will comply with the requirements of the protocol .
* Healthy subjects as established by medical history and physical examination.
* Access to a consistent means of telephone contact.
* For subjects who undergo a screening visit: results of all safety laboratory tests obtained at the screening visit must be within reference ranges. Results of any repeat testing cannot be used to qualify a subject for enrolment.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if they

  * have practiced adequate contraception for 30 days prior to vaccination, and
  * have a negative pregnancy test on the day of vaccination, and
  * agree to continue to practice adequate contraception until 2 months after the last dose administered.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence or evidence of substance abuse.
* Diagnosed with cancer, or treatment for cancer within three years.
* Diagnosed with excessive daytime sleepiness, or narcolepsy; or history of narcolepsy in a subject's parent, sibling or child.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 30 days prior to the first dose of study vaccine/placebo, or any other cytotoxic, immunosuppressive or immune-modifying drugs within 6 months of first study vaccine/ placebo dose.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine/placebo.
* Planned administration of any vaccine other than the study vaccine/placebo before blood sampling at the Day 42 visit.
* Previous administration of any H7 vaccine or physician-confirmed H7 disease.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within 90 days before the first dose of study vaccine/placebo, or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result before the first dose of study vaccine/placebo.
* Lactating or nursing women.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 424 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2015-01-19 (Actual)

PRIMARY OUTCOMES:
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers | At Day 42
  The following aggregate variables will be calculated for each adjuvanted H7N9 vaccine group: • Seroconversion rates (SCR); • Seroprotection rates (SPR); • Mean Geometric Increase (MGI)
Occurrence of each solicited local symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination
Occurrence of each solicited general symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination
Occurrence of clinical safety laboratory abnormalities reported for samples | At Day 0 visit
Occurrence of clinical safety laboratory abnormalities reported for samples | At Day 7 visit
Occurrence of clinical safety laboratory abnormalities reported for samples | At Day 21 visit
Occurrence of clinical safety laboratory abnormalities reported for samples | At Day 28 visit
Occurrence of clinical safety laboratory abnormalities reported for samples | At Day 42 visit
Occurrence of unsolicited adverse events | 21 days after each dose
Occurrence of Medically Attended Adverse Events (MAEs), potential Immune Mediated Diseases (pIMDs) and Serious Adverse Events (SAEs) | From Day 0 until the Day 42

SECONDARY OUTCOMES:
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers | At Day 42
  The following aggregate variables will be calculated for each adjuvanted (GSK3206641A) vaccine group which successfully meets CBER and CHMP criteria, and for the unadjuvanted (GSK3206640A) plain antigen vaccine group: • Geometric mean reciprocal serum HI antibody titers (GMTs); • SCR
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers | At Day 42
  The following aggregate variables will be calculated for the unadjuvanted plain antigen vaccine group: • SCR; • SPR; • MGI
Humoral immune response in terms of vaccine-homologous (H7N9) HI antibody titers | GMTs and Seropositivity rates at Days 0, 21, 42 and Months 6 and 12; SCR and MGI at Day 21, 42 (Placebo group only) and Months 6 and 12; SPR at Days 0, 21, 42 (Placebo group only) and Months 6 and 12
  The following aggregate variables will be calculated for each study group: • GMTs; • Seropositivity rates; • SCR; • SPR; • MGI
Humoral immune response in terms of vaccine-homologous (H7N9) HI antibody titers by age stratum | GMTs, Seropositivity rates and SPR at Days 0, 21, 42 and Months 6 and 12; SCR and MGI at Day 21, 42 and Months 6 and 12
  The following aggregate variables will be calculated for each study group by age stratum (18-40 years; 41-64 years): • GMTs; • Seropositivity rates; • SCR; • SPR; • MGI
Humoral immune response in terms of vaccine homologous (H7N9) neutralizing (MN) antibody titers | GMTs and Seropositivity rates at Days 0, 21, 42 and Month 6; VRR at Days 21, 42 and Month 6
  The following parameters will be calculated for a subset of subjects in each study group: • GMTs; • Seropositivity rates; • Vaccine response rate (VRR)
Occurrence of MAEs, pIMDs and SAEs | Until the Month 12 visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Seattle, Washington
- Canada (3):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Madan A, Segall N, Ferguson M, Frenette L, Kroll R, Friel D, Soni J, Li P, Innis BL, Schuind A. Immunogenicity and Safety of an AS03-Adjuvanted H7N9 Pandemic Influenza Vaccine in a Randomized Trial in Healthy Adults. J Infect Dis. 2016 Dec 1;214(11):1717-1727. doi: 10.1093/infdis/jiw414. Epub 2016 Sep 7. PMID 27609809
- See also: Results for study 201072 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/201072?search=study&#rs
- Available data/document: Informed Consent Form: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201072 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register